CLINICAL TRIAL: NCT04095559
Title: Characterization of Left Atrial Substrate by Comparison of Bipolar Voltage Maps With Standard Focal 4.5 mm Tip Electrode, 1 mm Ring Electrode, and Microelectrode Catheters Using InTEllaMap Orion and IntellaNav MIFI O
Acronym: CHAZESubstrate
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-01196; me19Kuehne2
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Atrial Fibrillation (AF)
Keywords: left atrial (LA) substrate-based ablation; focal ablation catheter; bipolar voltage amplitude; micro-electrode catheter; IntellaMap Orion; IntellaNav MIFI OI; bipolar voltage maps; irrigated-tip ablation catheter; ring-electrode circular mapping catheter; microelectrode multipolar catheter
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: multipolar mapping catheter — mapping of the left atrium will be performed in sinus rhythm using the IntellaMap Orion multipolar mapping catheter (Boston Scientific).
Diagnostic Test: multielectrode circular catheter — mapping of the left atrium will be performed using the multielectrode circular catheter (Lasso, spacing 2-6-2 mm, Biosense Webster)
Diagnostic Test: irrigated ablation catheter — mapping of the left atrium will be performed using the irrigated ablation catheter (IntellaNav Mifi OI)

SUMMARY:
This study is to investigate the correlation and to obtain the coefficient of correlation between the global and local bipolar signals (voltage maps) of the LA in sinus rhythm using a focal 4.5 mm irrigated-tip ablation catheter (in combination with microelectrodes), a ring-electrode circular mapping catheter and a microelectrode multipolar catheter in combination with the Rhythmia system.

DETAILED DESCRIPTION:
Current hypothesis of the mechanism of atrial fibrillation (AF) is a combination of local firing mainly triggered from the pulmonary veins and atrial substrate due to atrial remodelling sustaining AF. Whereas for paroxysmal AF, pulmonary vein isolation (PVI) is still the mainstay of interventional treatment, a left atrial (LA) substrate-based ablation especially in patients with persistent or long-standing persistent AF may be reasonable to improve freedom from AF. In addition, even in patients with paroxysmal AF, substrate-based ablation strategies have been shown to improve outcome. Substrate characterization of the LA is currently performed using the focal ablation catheter with a 3.5mm irrigated tip catheter with a 2 mm interelectrode spacing, a circular (Lasso) or spider like diagnostic (Pentaray) catheter with 1 mm size of the ring electrodes and 2 mm to 4 mm interelectrode spacing. Consequently, the cut-off values to delineate healthy tissue from diseased substrate are defined based on these measures. Since the electrode size and distance between the electrodes determines the bipolar voltage amplitude and morphology (beside their orientation with regard to the propagation wavefront), differences in bipolar voltage values must be expected between different catheter types and especially for the novel micro-electrode catheters IntellaMap Orion and IntellaNav MIFI OI. With the knowledge of the relationship between the bipolar voltage maps created with the different catheter types, information/knowledge from one study obtained with a specific catheter can be transferred to patients treated with the other catheter types. This study is to investigate the correlation and to obtain the coefficient of correlation between the global and local bipolar signals (voltage maps) of the LA in sinus rhythm using a focal 4.5 mm irrigated-tip ablation catheter (in combination with microelectrodes), a ring-electrode circular mapping catheter and a microelectrode multipolar catheter in combination with the Rhythmia system.

ELIGIBILITY:
Inclusion Criteria:

* Documented atrial fibrillation
* First or repeat catheter ablation

Exclusion Criteria:

* Previous heart surgery (high probability for atypical atrial tachycardia and non PV triggers for AF)
* Congenital heart disease (corrected or uncorrected)
* Severe uncorrected valvular heart disease
* Not willing or qualified for Magnetic Resonance Imaging of the heart
* Unable to provide informed consent
* Pregnancy (Pregnancy test will be performed before study participation)
* Patients with pacemaker or intracardiac defibrillator implanted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing catheter ablation for atrial fibrillation at the University Hospital Basel
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Global bipolar and unipolar signal measured in millivolt (mV) | single time point assessment at baseline
  Global bipolar and unipolar signal for the different types of catheters measured in mV
Local bipolar and unipolar signal measured in mV | single time point assessment at baseline
  Local bipolar and unipolar signal for the different types of catheters measured in mV

SECONDARY OUTCOMES:
Global fibrosis content and distribution from LGE-MRI measured in [%]. | single time point assessment at baseline
  Global fibrosis content and distribution from LGE-MRI measured in [%].
Local fibrosis content and distribution from Late-gadolinium enhanced Magnetic Resonance Imaging (LGE-MRI) measured in [%]. | single time point assessment at baseline
  Local fibrosis content and distribution from LGE-MRI measured in [%].
Differences of bipolar voltage characteristics between nearfield and farfield signals: amplitude (mV) | single time point assessment at baseline
  Differences of bipolar voltage characteristics between nearfield and farfield signals: amplitude (mV)
Differences of bipolar voltage characteristics between nearfield and farfield signals: frequency in Hertz (Hz) | single time point assessment at baseline
  Differences of bipolar voltage characteristics between nearfield and farfield signals: frequency (Hz)
Differences of bipolar voltage characteristics between nearfield and farfield signals: Duration in milliseconds (ms) | single time point assessment at baseline
  Differences of bipolar voltage characteristics between nearfield and farfield signals: duration (ms)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kuehne, Prof. Dr., Principal Investigator — Cardiology/Electrophysiology, University Hospital Basel
Locations (1):
- Cardiology/Electrophysiology, University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Schlageter V, Luca A, Badertscher P, Krisai P, Kueffer T, Spreen D, Katic J, Osswald S, Schaer B, Sticherling C, Kuhne M, Knecht S. Effect of electrode size and distance to tissue on unipolar and bipolar voltage electrograms and their implications for a near-field cutoff. Sci Rep. 2024 Nov 8;14(1):27184. doi: 10.1038/s41598-024-78627-5. PMID 39516302